CLINICAL TRIAL: NCT00700531
Title: European Trial of Free Light Chain Removal by Extended Haemodialysis in Cast Nephropathy
Acronym: EuLITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Birmingham (Other)
Collaborators: Gambro Renal Products, Inc. (Industry); Ortho Biotech, Inc. (Industry)
Responsible Party: Principal Investigator, Paul Cockwell, Doctor Paul Cockwell, University Hospital Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2007-003968-22; ISRCTN45967602
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Myeloma; Cast Nephropathy; Kidney Failure
Keywords: Hemodialysis; Multiple myeloma; Cast nephropathy; Kidney failure
MeSH Terms: conditions — Multiple Myeloma; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive FLC removal HD undertaken using an extended dialysis schedule on the Gambro HCO 1100 dialysers
  Interventions: Device: FLC removal HD (Gambro HCO 1100)
- 2 (Active Comparator): Patients receive standard dialysis on a high flux ployflux dialyser at a frequency determined by the duty nephrologist
  Interventions: Procedure: Standard dialysis on a high flux ployflux dialyser

INTERVENTIONS:
Device: FLC removal HD (Gambro HCO 1100) — FLC removal HD using a extended dialysis schedule on the Gambro HCO 1100
  Other Names: Gambro HCO 1100
  Arms: 1
Procedure: Standard dialysis on a high flux ployflux dialyser — Standard dialysis on a high flux ployflux dialyser at a frequency determined by the duty nephrologist
  Arms: 2

SUMMARY:
Hypothesis: Free light chain removal haemodialysis will increase the rate of renal recovery in patients with cast nephropathy, severe renal failure and de novo multiple myeloma.

This study will randomise patients with multiple myeloma and severe renal failure to treatment to remove free light chains by haemodialysis or not.

DETAILED DESCRIPTION:
The EUropean trial of free LIght chain removal by exTEnded haemodialysis in cast nephropathy (EuLITE) trial is a prospective, randomised, multicentre, open label clinical trial to investigate the clinical benefit of FLC removal haemodialysis in patients with cast nephropathy, dialysis dependent renal failure and de novo multiple myeloma. Recruitment commenced in May 2008, in total 90 patients will be recruited. Participants will be randomised, centrally, upon enrolment, to either trial chemotherapy and FLC removal haemodialysis or trial chemotherapy and standard high flux haemodialysis. Trial chemotherapy is a modified PAD regime, consisting of bortezomib, doxorubicin and dexamethasone. FLC removal haemodialysis is undertaken using two Gambro HCO 1100 dialysers in series, over an intensive treatment schedule. The primary outcome for the study is independence of dialysis at 3 months. Secondary outcomes are: duration of dialysis, reduction in serum FLC concentrations; myeloma response and survival.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Dialysis dependent acute renal failure (eGFR <15ml/min/1.73m2)
* Fulfils diagnostic criteria for the diagnosis of symptomatic de novo multiple myeloma1
* Abnormal serum FLC ratio and a sFLC concentration > 500 mg/L
* Myeloma kidney demonstrated on a renal biopsy (cast nephropathy)
* Ability to give informed consent to partake in study
* Commencement of study within 10 days of presenting to enrolling unit

Exclusion Criteria:

* Age < 18 years
* Known advanced chronic renal failure (CKD stage IV 4-5; eGFR <30mls/min/1.73m2) or evidence of significant chronic damage on renal biopsy
* Amyloidosis or light chain deposition disease on renal biopsy
* Previous treatment of multiple myeloma with chemotherapy
* Haemodynamic instability that precludes unsupported dialysis renal replacement therapy
* Significant cardiac disease (myocardial infarction with in the last 6 months; unstable angina; NYHA class III or IV heart failure; clinically significant pericardial disease; cardiac amyloidosis)
* Advanced disease or significant co-morbidity: with poor short term prognosis, necessitating palliation and no active or disease specific treatment.
* Inability to give informed consent
* History of allergic reaction attributable to compounds containing boron or mannitol
* History of Peripheral neuropathy or neuropathic pain (grade 2 or higher as defined by NCI CTCAE version 3)
* Clinically significant liver dysfunction (bilirubin >1.8mg/dl (30µmol/L))
* Known HIV infection
* Active uncontrolled infection
* Pregnant and lactating women
* Inability to give informed consent
* Pre-menopausal female patients of childbearing potential: positive pregnancy test or unwilling to use effective contraception during the study
* Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-06; Primary Completion 2014-01 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Independence of haemodialysis at 3 months from enrollment (eGFR > 15mls/min/1.73m2 at 2 weeks after last dialysis session) | 3 months from enrollment

SECONDARY OUTCOMES:
Efficiency of extended HD with respect to reduced sFLC concentrations; duration of HD before renal recovery; multiple myeloma response to chemotherapy and suitability for stem cell transplantation; mortality over 24 months observation period | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cockwell, PhD FRCP, Principal Investigator — University Hospital Birmingham; Mark Cook, PhD FRCPath, Principal Investigator — University Hospital Birmingham
Locations (1):
- University Hospital Birmingham, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Under consideration

REFERENCES:
- [Background] Hutchison CA, Cockwell P, Reid S, Chandler K, Mead GP, Harrison J, Hattersley J, Evans ND, Chappell MJ, Cook M, Goehl H, Storr M, Bradwell AR. Efficient removal of immunoglobulin free light chains by hemodialysis for multiple myeloma: in vitro and in vivo studies. J Am Soc Nephrol. 2007 Mar;18(3):886-95. doi: 10.1681/ASN.2006080821. Epub 2007 Jan 17. PMID 17229909
- [Background] Hutchison CA, Harding S, Mead G, Goehl H, Storr M, Bradwell A, Cockwell P. Serum free-light chain removal by high cutoff hemodialysis: optimizing removal and supportive care. Artif Organs. 2008 Dec;32(12):910-7. doi: 10.1111/j.1525-1594.2008.00653.x. PMID 19133018
- [Background] Hutchison CA, Cook M, Heyne N, Weisel K, Billingham L, Bradwell A, Cockwell P. European trial of free light chain removal by extended haemodialysis in cast nephropathy (EuLITE): a randomised control trial. Trials. 2008 Sep 28;9:55. doi: 10.1186/1745-6215-9-55. PMID 18822172